CLINICAL TRIAL: NCT05299411
Title: Preventive Effect of Intravenous Iron Infusion on Chemotherapy-induced Anemia of Colon Cancer Patients
Brief Title: Intravenous Iron Infusion on Chemotherapy-induced Anemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Pharmbio Korea Inc. (Unknown)
Responsible Party: Principal Investigator, Bong, Jun Woo, Clinical Associate Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021GR0540
Record Dates: First submitted 2022-03-10; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Colon Cancer; Chemotherapeutic-Induced Anemia
MeSH Terms: conditions — Colonic Neoplasms | interventions — iron isomaltoside 1000

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVI (Experimental): patients group with intravenous iron infusion
  Interventions: Drug: iron (isomaltoside)
- OI (Active Comparator): patients group with oral iron supplement
  Interventions: Drug: Dried Ferrous Sulfate

INTERVENTIONS:
Drug: iron (isomaltoside) — iron supplement through intravenous infusion
  Arms: IVI
Drug: Dried Ferrous Sulfate — iron supplement through oral intake
  Arms: OI

SUMMARY:
FOLFOX, the first-line regimen based on 5-FU and oxaliplatin, is adjuvant chemotherapy for pathologic stage II/III colorectal cancer patients. Among various side effects of FOLFOX, chemotherapy-induced anemia occurs in about 30% of patients with FOLFOX chemotherapy. An oral iron supplement is a widely accepted treatment for chemotherapy-induced anemia, but an oral iron supplement has a lot of inconveniences that can make patients' adherence worse, such as gastrointestinal discomfort, a long period of oral intake, and late recovery of serum iron level.

Intravenous iron infusion has been recently reported to be effective and safe to correct anemia. Previous studies reported that intravenous iron is also effective to correct chemotherapy-induced anemia. However, there is a paucity of studies associated with colorectal cancer patients with FOLFOX chemotherapy.

This study aimed to evaluate the effect of intravenous iron on chemotherapy-induced anemia after FOLFOX chemotherapy for patients with colorectal cancer compared with the effect of oral iron supplements. Parameters including serum Hb, serum iron, serum ferritin concentrations, total iron-binding capacity, absolute neutrophil count, platelet, albumin, C reactive protein, hepcidin, soluble transferrin receptor, and IL6 will be analyzed. In addition, information on chemotoxicity, adverse events during chemotherapy and quality of life will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* * clinical diagnosis of stage II or III after curative resection for colon cancer and planned to be received modified FOLFOX6 as an adjuvant chemotherapy

  * more than 18 years old
  * baseline Hb level <12g/dL or more Hb 2g/dL decrease after chemotherapy
  * patients who received more than 1 cycle of FOLFOX6

Exclusion Criteria:

* * patients with neoadjuvant therapy

  * patients who have other diseases associated with anemia such as CKD, IBD, other bone marrow diseases
  * patients who received RBC transfusion during chemotherapy
  * patients diagnosed with local recurrence or distant metastasis during chemotherapy
  * ferritin > 800 ng/mL and TSAT ≧ 50%
  * patients who are not willing to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum Hb level | during chemotherapy

SECONDARY OUTCOMES:
Serum hepcidin level | during chemotherapy

OTHER OUTCOMES:
Quality of life associated anemia | during chemotherapy
  FACT-An (Version 4)